CLINICAL TRIAL: NCT02194543
Title: High-Definition 3D Visualization System for Ophthalmic Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2014-0002
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Cataract
Keywords: Cataract; HD 3D; Microscope
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HD 3D: The patients received surgeries with HD 3D on their left eyes.
- Conventional: The patients received surgeries with conventional method on the other eye.

SUMMARY:
To validate a high-definition (HD) three-dimensional (3D) visualization system in cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* The patients are scheduled to cataract surgery on both eyes.

Exclusion Criteria:

* The patients who have other complicating ophthalmic diseases or previous history of ophthalmic surgeries were excluded

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cataract
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
the best corrected visual acuity | 1 month after the operation
  operation time, total phacoemulsification time, and postoperative visual outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea